CLINICAL TRIAL: NCT01803932
Title: Evaluation of a Male-focused Primary Prevention Intervention to Prevent Intimate Partner Violence in a Conflict-affected Setting: A Cluster Randomized Controlled Trial in Cote d'Ivoire
Brief Title: Evaluation of a Male-focused Intervention to Prevent Intimate Partner Violence in a Conflict-affected Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: International Rescue Committee (Other)
Responsible Party: Principal Investigator, Mazeda Hossain, Principal Investigator, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: InterveneDV-CI
Record Dates: First submitted 2013-02-25; First posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Domestic Violence
Keywords: intimate partner violence; gender; primary prevention intervention; conflict; Cote d'Ivoire; Ivory Coast
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral intervention (Experimental): Male-focused group violence prevention intervention
  Interventions: Behavioral: Male-focused group violence prevention intervention
- Control communities (No Intervention): Communities in which male-focused group prevention activities will not be conducted

INTERVENTIONS:
Behavioral: Male-focused group violence prevention intervention
  Arms: Behavioral intervention

SUMMARY:
Cluster randomized controlled trial to evaluate a male-focused primary prevention programme which used a men's only group discussion format to prevent intimate partner violence against women & girls through fostering knowledge and behaviour changes by: (1) increasing men's knowledge on the impact of violence against women; (2) promoting gender equitable beliefs/behaviours within relationships; and (3) developing anger management techniques.

ELIGIBILITY:
Inclusion Criteria:

* 15+ years old
* males: participant in group intervention or selected as control
* females: female intimate partner of males in intervention or selected as control
* capable of completing face-to-face interview independently and without causing undue psychological distress

Exclusion Criteria:

* lack of informed consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Past 12 months victimisation/perpetration of physical or sexual intimate partner violence | 1 year after intervention completion

CONTACTS AND LOCATIONS:
Overall Officials: Mazeda Hossain, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- International Rescue Committee, Abidjan, Côte d’Ivoire

REFERENCES:
- [Derived] Hossain M, Zimmerman C, Kiss L, Abramsky T, Kone D, Bakayoko-Topolska M, Annan J, Lehmann H, Watts C. Working with men to prevent intimate partner violence in a conflict-affected setting: a pilot cluster randomized controlled trial in rural Cote d'Ivoire. BMC Public Health. 2014 Apr 10;14:339. doi: 10.1186/1471-2458-14-339. PMID 24716478